CLINICAL TRIAL: NCT04038762
Title: Tracheal Tube Cuff Inflation-deflation Method for Video Laryngoscope-assisted Nasal Intubation in Pediatric Patients
Brief Title: Inflation-deflation Method for Nasal Intubation in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Tarek F.Tammam, Tarek F.Tammam,M.D,Ph.D,Department of Anesthesia and intendive care,Faculty of Medicine., Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Tammam
Record Dates: First submitted 2019-07-22; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Nasal Intubation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional nasal intubation (Active Comparator): Passage of an endotracheal tube via the nare followed by video laryngoscopy-assisted passage through the glottis, with or without the aid of Magill forceps
  Interventions: Procedure: cuff deflation-inflation -deflation method
- Nasotracheal Intubation with cuff inflation-deflation method (Experimental): Nasotracheal intubation placed with video laryngoscopy assistance, via the tracheal tube cuff inflation-deflation method with or without the aid of Magill forceps
  Interventions: Procedure: cuff deflation-inflation -deflation method

INTERVENTIONS:
Procedure: cuff deflation-inflation -deflation method — Nasotracheal intubation placed with video-laryngoscopy assistance, via the tracheal tube cuff inflation-deflation method with or without the aid of Magill forceps
  Other Names: pre-cuff inflation

SUMMARY:
Magill forceps is used to maneuver the endotracheal tube ETT in the posterior oropharynx and place its tip into the laryngeal inlet. While the Magill forceps are useful in guiding the nasotracheal tube past the vocal cords, care must be taken to avoid excessive maneuvering in order to minimize the risk of local trauma and rupture of the nasotracheal tube balloon.

Cuff inflation-deflation method can reduce the apnea time in the pediatric patients, a population with known physiological limitations in respiratory reserve. This, in turn, could point to a reduction in the complications (as desaturation and cardiac arrhythmia) that associated with the prolonged-time procedure.

DETAILED DESCRIPTION:
the investigator will compare the cuff inflation-deflation method versus the conventional method of nasal intubation in pediatric patients for the need of using Magill forceps 90 pediatric patients between the ages of 3 and 12 years with the American Society of Anesthesiologists (ASA) physical status I-II, scheduled for elective surgery (dental and maxillofacial) will be enrolled in a prospectively randomized observer-blinded clinical trial. Patients, who have coagulopathies, have upper airway abnormalities, at risk for aspiration or by reasons of parent's refusal will be excluded from the study.

Airway management is subdivided into phases:

* Phase 1: Passage of the endotracheal tube through the nose into the pharynx
* Phase 2: Video-laryngoscope-guided passage of the endotracheal tube through the pharynx into the trachea.

Phase 2 can be performed with the tracheal tube cuff inflation-deflation method vs. non-cuff inflation method. A Magill forceps can be used to guide the endotracheal tube pass through the pharynx and glottis into the trachea if required.

Tracheal tube cuff inflation-deflation method: Tracheal tube cuff is inflated with a variable amount of air (volume of air is depending on the level of the larynx). Once the tip of endotracheal tube at the laryngeal inlet, the cuff of the endotracheal tube is deflated and advanced into the trachea

Patients included in the study will be assigned into two groups for the second phase of airway management:

Group A (n = 45) in whom nasal intubation will be performed using the cuff inflation-deflation method; and Group B (n = 45), in whom the nasal intubation will be performed using non-inflation method.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II,
* Scheduled for elective surgery (dental and maxillofacial) in need for nasal intubation.

Exclusion Criteria:

* Patients, who have coagulopathies,
* Have upper airway abnormalities,
* At risk for aspiration or by reasons of
* Parent's refusal will be excluded from the study

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
to test whether the inflation-deflation method (pre-cuff inflation) would decrease the need for Magill forceps in video laryngoscopy assisted nasal intubation in pediatric patients compared with the conventional non-cuff inflation approach. T | during nasal intubation : 60 seconds
  The percentage of patients who did not require Magill forceps for nasal intubation success was recorded.

SECONDARY OUTCOMES:
The time period for the second phase nasal intubation | 60 seconds
  The time in seconds for the second phase nasal intubation
The number of attempts required for successful nasal intubation. | 120 seconds
  number of trials, how many numbers of attempts the investigator take for successful nasal intubation
Amount of injected air for cuff inflation | 15 seconds
  Amount of injected air in ml, how many air injected in the cuff balloon to make the tip of endotracheal tube advanced into the trachea
Assessment of side effects of using Magill forceps during nasal intubation | Intraoperative and in the first 48 postoperative hours]
  A 4-point scale: 1- No epistaxis; 2-Mild epistaxis (blood on the tracheal tube only); 3- Moderate epistaxis (blood pooling in the pharynx); 4- Severe epistaxis (blood in the pharynx sufficient to impede intubation)
Evaluation of oxygenation state during nasal intubation | preoperative and intraoperative
  rate of oxygen drop during the procedure
evaluate the anesthetists' experience of using the inflation-deflation method for nasal intubation. | 20 minutes after complete recovery of patients
  score 1 to 5 A five-point Likert scales for: How likely is it that anesthetist would recommend the same used inflation-deflation method to practice a colleague in the future (not at all/ slightly/ moderately/ very/ extremely: where 1 is not at all, 3 is moderate,5 is extremely

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek F.Tammam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No